CLINICAL TRIAL: NCT00621010
Title: A Phase 1 Single Escalating Dose Study to Assess the Safety and Pharmacokinetics of CTS21166 Administered Intravenously to Healthy Adult Males
Brief Title: Safety Study of CTS21166 to Treat Alzheimer Disease
Acronym: CTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CoMentis (Industry)
Responsible Party: Henry Hsu, MD, Comentis, Inc.
Purpose: Treatment
Other Study IDs: CTS21166-101
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: CTS21166 (ZPQ-21166)

INTERVENTIONS:
Drug: CTS21166 (ZPQ-21166) — Cohort 1: (7.5 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days; Cohort 2: (22.5 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days; Cohort 3: (45 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days; Cohort 4: (90 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days; Cohort 5: (150 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days; Cohort 6: (225 mg): 6 subjects, plus 2 placebo. If no safety concerns after 7 days,proceed to Part B.
  Cohort 7: (225 mg): Up to 10 subjects, open label, 3 hour infusion

SUMMARY:
This study is the first human exposure for the drug candidate CTS21166 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male > age 21;
* non-smoker (minimum 6 months);

Exclusion Criteria:

* History or evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic,neurologic, psychiatric, oncologic, or allergic (including anaphylactic drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease
* History or evidence of intravenous illicit drug use, human immunodeficiency virus (HIV), hepatitis B, or hepatitis C;
* Participation in another clinical trial within 30 days prior to dosing

Min Age: 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending doses of CTS21166 following intravenous administration

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics(PK) of CTS21166 and its major metabolites as assessed in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, M.D., Study Director — CoMentis
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States